CLINICAL TRIAL: NCT01102283
Title: Treatment of Colonic Obstruction With Cook Evolution® Colonic Stent System
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-022; 100041 (Other: Cook)
Record Dates: First submitted 2010-03-29; First posted 2010-04-13 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Colonic Obstruction; Colonic Stricture; Large Bowel Obstruction
Keywords: Colonic obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Stent Group
  Interventions: Device: Evolution(R) Colonic Stent

INTERVENTIONS:
Device: Evolution(R) Colonic Stent — Palliative treatment of colonic obstruction or strictures caused by malignant neoplasms and to relieve acute large bowel obstruction prior to colectomy in patients with malignant strictures.

SUMMARY:
The objective of this registry is to compile clinical data on the use of the Evolution® Colonic Stent System for the palliative treatment of colonic obstruction or strictures caused by malignant neoplasms and to relieve acute large bowel obstruction prior to colectomy in patients with malignant strictures.

ELIGIBILITY:
Inclusion: per the IFU,

* colonic strictures caused by malignant neoplasms, and
* large bowel obstruction due to malignant strictures prior to colectomy.

Exclusion:

* central ischemia,
* any contraindication to GI endoscopy and any procedure to be performed in conjunction with stent placement,
* suspected or impending perforation,
* intra-abdominal abscess/perforation,
* inability to pass wire guide or stent deployment system through the obstructed area,
* patients for whom endoscopic or percutaneous procedures are contraindicated,
* benign disease, and
* coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Referral Centers
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Relief of obstruction | At the Conclusion of the Procedure

SECONDARY OUTCOMES:
Implant Duration | 6 months
Symptoms at Follow-up | 6 months
Complications | 6 months
  perforation, migration, obstruction, GI bleeding requiring intervention

CONTACTS AND LOCATIONS:
Locations (10):
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Odense Universitetshospital, Odense, Denmark
- Institut Paoli Calmettes, Marseille, France
- Instituto Clinico Humanitas IRCCS, Milan, Italy
- Deventer Ziekenhuis, Deventer, Netherlands
- Spain (3):
  - Hospital de Basurto, Bilbao, Bilbao
  - Hospital Universitari de Girona, Girona
  - Hospital Son Llatzer, Palma de Mallorca
- University College of London Hospital, London, United Kingdom